CLINICAL TRIAL: NCT02144454
Title: The Acute Effects of Meals Rich in Saturated, Monounsaturated and n-6 Polyunsaturated Fatty Acids on Vascular Function
Brief Title: Impact of Meal Fatty Acids on Postprandial Vascular Reactivity
Acronym: DIVAS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Department of Health, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor Julie Lovegrove, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 024/0036
Record Dates: First submitted 2014-05-15; First posted 2014-05-22 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Fatty acids; Vascular function; Blood pressure; Plasma lipids; Insulin resistance; Endothelial activation
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance | interventions — Fatty Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Meal rich in saturated fats (Active Comparator): Subjects are asked to consume a breakfast (0 min) and lunch (330 min) rich in saturated fats
  Interventions: Dietary Supplement: Saturated fat
- Meal rich in monounsaturated fats (Experimental): Subjects are asked to consume a breakfast (0 min) and lunch (330 min) rich in monounsaturated fats
  Interventions: Dietary Supplement: Monounsaturated fat
- Meal rich in n-6 polyunsaturated fats (Experimental): Subjects are asked to consume a breakfast (0 min) and lunch (330 min) rich in n-6 polyunsaturated fats
  Interventions: Dietary Supplement: n-6 polyunsaturated fat

INTERVENTIONS:
Dietary Supplement: Saturated fat
  Other Names: SFA
  Arms: Meal rich in saturated fats
Dietary Supplement: Monounsaturated fat
  Other Names: MUFA
  Arms: Meal rich in monounsaturated fats
Dietary Supplement: n-6 polyunsaturated fat
  Other Names: n-6 PUFA
  Arms: Meal rich in n-6 polyunsaturated fats

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in women. Premenopausal women have a lower risk of CVD compared with men of a similar age. However, the incidence of CVD increases greatly after the menopause. The risk of heart disease is strongly associated with the health of an individual's blood vessels. It is thought that changes to the type of fat the investigators eat in their diet may affect the normal functioning and elasticity of the blood vessels, as well as affect cholesterol levels in the blood. Types of fat in the diet include monounsaturated fats (found mainly in olive oil), n-6 polyunsaturated fats (found mainly in sunflower oil) and saturated fats (found mainly in dairy products, such as butter and cheese). Since the investigators are in the fed (or postprandial) state for up to 18 hours of the day, it is important to see how these different fats affect the investigators blood vessels and blood fats over the course of the day after eating a meal. The aim of this study is to determine how consuming meals rich in saturated fats, n-6 polyunsaturated fats or monounsaturated fats influence the normal functioning and elasticity of the blood vessels throughout the day in postmenopausal women. A secondary aim is to determine the effects of these different dietary fats on a range of accepted heart disease risk markers including circulating levels of fats (lipids) and glucose in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (not menstruated for at least 1 year)
* Plasma triacylglycerol (TAG) between 0.8 and 4.0 mmol/l
* Body mass index (BMI) between 18-35 kg/m2
* Total cholesterol (TC): <8 mmol/l
* Systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg
* Non-smoker

Exclusion Criteria:

* Having suffered a myocardial infarction/stroke in the past 12 months
* Diabetic (diagnosed as fasting blood glucose >7 mmol/l) or suffering from other endocrine disorders
* Suffering from renal or bowel disease or have a history of cholestatic liver or pancreatitis
* On drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* History of alcohol abuse
* On hormone replacement therapy (HRT)
* Planning or on a weight reducing regime
* Taking nutritional supplements (e.g. fish oil, calcium)
* Anaemic: haemoglobin <11.5 g/dl

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vascular reactivity measured by flow-mediated dilatation (FMD) | Acute study: measured at 0 (baseline), 180, 300 and 420 min

SECONDARY OUTCOMES:
Change from baseline in vascular reactivity measured by laser Doppler imaging with iontophoresis of acetylcholine (endothelium-dependent) and sodium nitroprusside (endothelium-independent) | Acute study: measured at 0 (baseline), 240 and 450 min
Change from baseline in plasma lipids (primarily triacylglycerol, apolipoprotein B and non-esterified fatty acids) | Acute study: taken at 30 min intervals between 0 min (baseline) and 480 min
Change from baseline in arterial stiffness measured by digital volume pulse (stiffness index and reflection index) | Acute study: taken at 0 (baseline), 240 amd 450 min
Change from baseline in blood pressure (systolic blood pressure, diastolic blood pressure and pulse pressure) | Acute study: taken at 0 (baseline), 240 and 450 min
Change from baseline in markers of insulin resistance (glucose, insulin, indices of insulin resistance/sensitivity) | Acute study: taken at 30 min intervals between 0 min (baseline) and 480 min
Change from baseline in nitric oxide (total plasma nitrates and nitrites) | Acute study: 0 (baseline), 180, 300 and 420 min
Change from baseline in plasma markers of endothelial activation (e.g. E-selectin, P-selectin, vascular cell adhesion molecule (VCAM-1)) | Acute study: 0 (baseline), 180, 300 and 420 min
Change from baseline in plasma phospholipid fatty acid composition | Acute study: 0 (baseline), 180, 300 and 420 min

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc PhD RNutr, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Rathnayake KM, Weech M, Lovegrove JA, Jackson KG. Glu298Asp (rs1799983) Polymorphism Influences Postprandial Vascular Reactivity and the Insulin Response to Meals of Varying Fat Composition in Postmenopausal Women: Findings from the Randomized, Controlled Dietary Intervention and VAScular function (DIVAS)-2 Study. J Nutr. 2021 Apr 8;151(4):848-856. doi: 10.1093/jn/nxaa394. PMID 33693945
- [Derived] Rathnayake KM, Weech M, Jackson KG, Lovegrove JA. Meal Fatty Acids Have Differential Effects on Postprandial Blood Pressure and Biomarkers of Endothelial Function but Not Vascular Reactivity in Postmenopausal Women in the Randomized Controlled Dietary Intervention and VAScular function (DIVAS)-2 Study. J Nutr. 2018 Mar 1;148(3):348-357. doi: 10.1093/jn/nxx042. PMID 29546297